CLINICAL TRIAL: NCT05467358
Title: The Effect of Using Preendoscopic Proton Pump Inhibitors in Upper Gastrointestinal System Bleeding on Patient Prognosis
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: AnkaraCHBilkent-nısık-002
Record Dates: First submitted 2022-06-17; First posted 2022-07-20 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2022-07

CONDITIONS: Upper Gastrointestinal Bleeding, Proton Pump Inhibitors
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with preendoscopic ppi order: Patients receiving 80 mg esomeprazole loading and 8 mg esomeprazole infusion per hour before endoscopic treatment
- Patients with preendoscopic cannot be ppi order: patients who could not get ppi before endoscopy

SUMMARY:
In this study, we aimed to investigate the effectiveness of ppi use in upper gastrointestinal bleeding in patients over the age of 18 who underwent endoscopy on mortality, length of hospital stay, rebleeding, and cost. The European Society of Gastrointestinal Endoscopy 2021 recommends the use of preendoscopic ppi in patients with nonvariceal upper gastrointestinal bleeding as it reduces the need for endoscopic treatment. This recommendation is recommended by the British Institute for Health and Care Excellence not to use proton pump inhibitors. Likewise, the 2021 American Gastroenterology Association did not make a recommendation for its use because the benefit of using preendoscopic ppi is uncertain. This has led to confusion about the efficacy of ppi and has questioned the necessity of routinely given high-dose ppi therapy. In this study, we aim to reveal the effectiveness of the treatment by comparing the patients who were given and not given ppi. Our research is a retrospective cohort study. Patients over the age of 18 who applied to the emergency department and had a preliminary diagnosis of upper gastrointestinal bleeding and underwent endoscopy will be included in the study. Patients who underwent endoscopy and were given ppi and those who were not will be compared. In upper gastrointestinal bleeding, patients with a Glasgow Blatchford score of 2 and above are taken to endoscopy. Therefore, patients over the age of 18 who underwent endoscopy will be included in the study.

DETAILED DESCRIPTION:
Due to the problems experienced in the supply of ppi, ppi was not available in our hospital for a while. Therefore, ppi could not be given to the patients. It was started to be given after the drug was re-supplied. In our study, we retrospectively analyzed patients who could and could not receive ppi. The data of the patients were as follows: age, gender, complaints on admission, known diseases, vital signs, medications used, rectal examination, whole blood parameters, biochemistry parameters, Glasgow Blatchford scores, endoscopy results, whether they received blood products, how much of each product they received, emergency We recorded service outcomes and emergency room costs.

ELIGIBILITY:
Inclusion Criteria:

* having an endoscopy at the time of admission to the emergency room
* Glasgow Blatchford score of 2 or higher
* be over 18 years old

Exclusion Criteria:

* patients who do not meet the inclusion criteria will be excluded

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients admitted to the emergency department with suspected upper gastrointestinal bleeding and undergoing endoscopy
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Need for repeat endoscopy | 7 days
  Bleeding associated need for reoperation
mortality | 28 days
  illness related death
hospital stay time | through study completion, an average of 1 year
  hospitalization day
cost of transactions | through study completion, an average of 1 year
  health expenditure during hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: GÜLHAN KURTOĞLU ÇELİK, Prof.Dr., Study Director — ANKARA CİTY HOSPİTAL
Locations (1):
- Ankara Bilkent Şehir Hastanesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Data can be shared if researchers who are considering making a meta-analysis on the subject contact.

REFERENCES:
- [Background] Daneshmend TK, Hawkey CJ, Langman MJ, Logan RF, Long RG, Walt RP. Omeprazole versus placebo for acute upper gastrointestinal bleeding: randomised double blind controlled trial. BMJ. 1992 Jan 18;304(6820):143-7. doi: 10.1136/bmj.304.6820.143. PMID 1737157
- [Background] Lau JY, Leung WK, Wu JC, Chan FK, Wong VW, Chiu PW, Lee VW, Lee KK, Cheung FK, Siu P, Ng EK, Sung JJ. Omeprazole before endoscopy in patients with gastrointestinal bleeding. N Engl J Med. 2007 Apr 19;356(16):1631-40. doi: 10.1056/NEJMoa065703. PMID 17442905
- [Background] Laine L, Barkun AN, Saltzman JR, Martel M, Leontiadis GI. ACG Clinical Guideline: Upper Gastrointestinal and Ulcer Bleeding. Am J Gastroenterol. 2021 May 1;116(5):899-917. doi: 10.14309/ajg.0000000000001245. PMID 33929377
- [Background] Gralnek IM, Stanley AJ, Morris AJ, Camus M, Lau J, Lanas A, Laursen SB, Radaelli F, Papanikolaou IS, Curdia Goncalves T, Dinis-Ribeiro M, Awadie H, Braun G, de Groot N, Udd M, Sanchez-Yague A, Neeman Z, van Hooft JE. Endoscopic diagnosis and management of nonvariceal upper gastrointestinal hemorrhage (NVUGIH): European Society of Gastrointestinal Endoscopy (ESGE) Guideline - Update 2021. Endoscopy. 2021 Mar;53(3):300-332. doi: 10.1055/a-1369-5274. Epub 2021 Feb 10. PMID 33567467
- [Background] Pouw RE, Barret M, Biermann K, Bisschops R, Czako L, Gecse KB, de Hertogh G, Hucl T, Iacucci M, Jansen M, Rutter M, Savarino E, Spaander MCW, Schmidt PT, Vieth M, Dinis-Ribeiro M, van Hooft JE. Endoscopic tissue sampling - Part 1: Upper gastrointestinal and hepatopancreatobiliary tracts. European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2021 Nov;53(11):1174-1188. doi: 10.1055/a-1611-5091. Epub 2021 Sep 17. PMID 34535035